CLINICAL TRIAL: NCT04435730
Title: Use of Serum Mac-2 Binding Protein and Musculoskeletal Ultrasound to Predict Arthritis in Psoriatic Patients
Brief Title: Use of Serum M2BP and MSUS to Predict Arthritis in Psoriatic Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sylvia Victor Anis Ross, Sylvia Victor, Assiut University
Other Study IDs: M2BP and MSUS in psoriasis
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: 45 patients with cutaneous psoriasis with no musculoskeletal manifestations.
  Interventions: Diagnostic Test: serum level of Mac 2 binding protein; Device: musculoskeletal ultrasound
- Group 2: 45 patients with psoriatic arthritis fulfilling CASPAR criteria of PsA
  Interventions: Diagnostic Test: serum level of Mac 2 binding protein; Device: musculoskeletal ultrasound
- Group 3: 45 patients with subclinical psoriatic arthritis (patients with cutaneous psoriasis and musculoskeletal manifestations but not fulfilling CASPARcriteria of PsA).
  Interventions: Diagnostic Test: serum level of Mac 2 binding protein; Device: musculoskeletal ultrasound
- Group 4: 45 sex and age matched healthy controls
  Interventions: Diagnostic Test: serum level of Mac 2 binding protein; Device: musculoskeletal ultrasound

INTERVENTIONS:
Diagnostic Test: serum level of Mac 2 binding protein — Serum levels of Mac 2 binding protein will be measured for all the study subjects using Enzyme-Linked Immuno sorbent Assay (ELISA).
  2 ml of venous blood will be collected from patients and controls under complete aseptic conditions in a plain tube. Sample will be allowed to clot for 15-30 min at room temperature and then centrifuged at 2500 rpm for 10-15 min. Serum will be separated and stored at -20 C or lower till time of assessment.
Device: musculoskeletal ultrasound — MSUS examination will be performed for patients of all groups and control group.Gray scale (GSUS) and power Doppler (PDUS) at joints levels and entheses will be performed with the same transducer of My Lab Seven Crystalline esaote machine.

SUMMARY:
Aims of the study:

1. Measurement of serum level of Mac 2 binding protein among patients with psoriasis, psoriatic arthritis and subclinical psoriatic arthritis compared with healthy individuals.
2. Evaluation of MSUS findings in patients with PsA and subclinical psoriatic arthritis
3. Evaluation of the role of serum level of Mac 2 binding protein and MSUS in predicting arthritis among psoriatic patients.

DETAILED DESCRIPTION:
Psoriasis is a quite common chronic, inflammatory immune-mediated skin disease affecting about 2% of the population . Also psoriasis is a strong risk factor for the development of several comorbidities of which the most common is psoriatic arthritis (PsA).

The presence of cutaneous psoriasis indicates a high risk for developing PsA. Studies conducted in dermatology clinics have shown a high prevalence of undiagnosed PsA in psoriasis patients , therefore identifying soluble biomarkers for PsA in psoriasis patients may help in early diagnosis, and thereby prevent disability and improve quality of life .

Mac 2 binding protein [M2BP] is thought to be a marker of synovial cell activation and joint destruction .M2BP may be involved in the pathogenesis of PsA .

Recently, with the introduction of new medications and wider use of musculoskeletal ultrasound (US) imaging in clinical practice, the possibility of earlier US diagnosis in patients with psoriasis in the pre-clinical phase of PsA has been examined.

ELIGIBILITY:
Inclusion Criteria:

cutaneous psoriasis Psoriatic arthritis Subclunical psoriatic arthritis

Exclusion Criteria:

any history of liver diseases non-alcoholic fatty liver, viral hepatitis, human immunodeficiency virus (HIV), autoimmune rheumatic disease other than psoriasis and PSA malignancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a case control, cross section study and will include patients with psoriasis, psoriatic arthritis, subclinical psoriatic arthritis and healthy controls aged > 18 years. .
  Patients involved in the research will be selected from both Dermatology and Rheumatology and Rehabilitation outpatient clinic and inpatient word in Assuit University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
measurement of serum level of M2BP among psoriasis , psoriatic arthritis and subclinical psoriatic arthritis patients compared with healthy individuals and evaluation of MSUS findings in patients with PsA and subclinical psoriatic arthritis | baseline
  detection of the role of serum level of Mac 2 binding protein and MSUS to predict arthritis among psoriatic patients

CONTACTS AND LOCATIONS:
Overall Officials: Safaa Mahran, Study Chair — Assiut University
Locations (1):
- Sylvia, Asyut, Egypt

REFERENCES:
- [Background] Ritchlin CT, Colbert RA, Gladman DD. Psoriatic Arthritis. N Engl J Med. 2017 Mar 9;376(10):957-970. doi: 10.1056/NEJMra1505557. No abstract available. PMID 28273019
- [Background] Cretu D, Gao L, Liang K, Soosaipillai A, Diamandis EP, Chandran V. Differentiating Psoriatic Arthritis From Psoriasis Without Psoriatic Arthritis Using Novel Serum Biomarkers. Arthritis Care Res (Hoboken). 2018 Mar;70(3):454-461. doi: 10.1002/acr.23298. PMID 28586166
- [Background] Cretu D, Prassas I, Saraon P, Batruch I, Gandhi R, Diamandis EP, Chandran V. Identification of psoriatic arthritis mediators in synovial fluid by quantitative mass spectrometry. Clin Proteomics. 2014 Jul 1;11(1):27. doi: 10.1186/1559-0275-11-27. eCollection 2014. PMID 25097465